CLINICAL TRIAL: NCT00436033
Title: A European Phase III, Multicentre, Double-blind, Randomised, Placebo-controlled Monotherapy Study of Milnacipran for the Treatment of Fibromyalgia Syndrome
Brief Title: A Multicentre Trial to Determine the Efficacy and Safety of Milnacipran in the Treatment of Fibromyalgia Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F02207GE302
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Minalcipran (Experimental)
  Interventions: Drug: milnacipran

INTERVENTIONS:
Drug: milnacipran
  Arms: Minalcipran
Drug: Placebo
  Arms: Placebo

SUMMARY:
Investigation of efficacy and safety of treatment with milnacipran in the treatment of fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patient with a diagnosis of fibromyalgia according to the 1990 American College of Rheumatology (ACR) criteria

Exclusion Criteria:

* psychiatric illness
* depression of generalised anxiety disorder
* suicidal risk
* substance abuse
* active cardiac disease
* pulmonary dysfunction
* liver disease
* renal impairment
* autoimmune disease
* chronic inflammatory rheumatoid disease
* current systemic infection
* epileptic
* active cancer
* sleep apnea
* active peptic ulcer
* inflammatory bowel disease
* unstable endocrine disease
* for men : prostatic enlargement of genito-urinary disorders
* for women : pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1429 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of treatment with milnacipran as compared to placebo in the treatment of the fibromyalgia syndrome in outpatients after a 12-week period of fixed dose exposure through a primary composite criterion | 12 weeks

SECONDARY OUTCOMES:
comparison of efficacy of treatment with milnacipran to placebo on additional secondary criteria | 12 weeks
establishment of safety profile of treatment of milnacipran in patients with fibromyalgia syndrome (FMS). | 19 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jaime C BRANCO, Principal Investigator — HOSPITAL EGAS MONIZ
Locations (13):
- Rheumatology Ambulance, Pardubice, Czechia
- FREDERIKSBERG HOSPITAL - Clinic of Rheumatology, Frederiksberg, Denmark
- Kuopion Oma Laakari Oy, Kuopio, Finland
- Hopital Hotel Dieu, Paris, France
- KKSK KLINIKUM DER UNIVERSITAET ZU KOELN - Anaesthesiology and Intensive Care, Cologne, Germany
- Ospedale Luigi Sacco, Milan, Italy
- Center For Clinical Studies, Lillehamer, Norway
- "Nasz Lekarz", Torun, Poland
- Hospital Egas Moniz, Lisbon, Portugal
- Dr I CANTACUZINO CLINICAL HOSPITAL, Bucharest, Romania
- Hospital de La Esperanza, Barcelona, Spain
- Gottfriesclinic Ab, Mölndal, Sweden
- KINGS COLLEGE HOSPITAL - Clinic Trial Unit Academic Department of Rheumatology, London, United Kingdom

REFERENCES:
- [Derived] Branco JC, Zachrisson O, Perrot S, Mainguy Y; Multinational Coordinator Study Group. A European multicenter randomized double-blind placebo-controlled monotherapy clinical trial of milnacipran in treatment of fibromyalgia. J Rheumatol. 2010 Apr;37(4):851-9. doi: 10.3899/jrheum.090884. Epub 2010 Feb 15. PMID 20156949